CLINICAL TRIAL: NCT04747665
Title: Patient and Endoscopists' Experiences and Perceptions of Colonoscopy and New Technologies in Colonoscopy
Brief Title: Experiences and Perceptions of Colonoscopy and New Technologies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 281674
Record Dates: First submitted 2021-01-27; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Bowel Cancer; Colonoscopy
Keywords: Endoscopy; Colonoscopy; Robotic colonoscopy; Artificial intelligence; Patient reported experience
MeSH Terms: conditions — Intestinal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients who have undergone or refused to undergo colonoscopy
  Interventions: Other: Patient and endoscopist reported experience
- Endoscopists: Endoscopists who perform or are training to perform colonoscopy
  Interventions: Other: Patient and endoscopist reported experience

INTERVENTIONS:
Other: Patient and endoscopist reported experience — Exploration of patient and endoscopists experiences of colonoscopy.

SUMMARY:
Bowel cancer is the 3rd most common cancer in males and females. Most bowel cancers develop from precancerous polyps in the bowel. Colonoscopy can detect and remove these polyps, thereby reducing the risk of developing bowel cancer. However, colonoscopy is an invasive procedure with inherent risk, and can be both uncomfortable and embarrassing to undergo. The risks and numerous other barriers often mean colonoscopy, and cancer preventing polyp removal, is not performed.

The investigators aim to start the first in-human feasibility clinical investigation of a robotic magnetic colonoscope in 2021. The new device aims to reduce the discomfort and risk associated with colonoscopy. As part of the patient and end user involvement aspect of the project the investigators aim to perform a mixed methodology inductive type research project exploring experiences of colonoscopy for patient and endoscopists.

The study will follow an exploratory mixed methodology format with two parallel work-streams for patients and endoscopists. Each work-stream will consisting of a focus groups (1-2 for each patients and endoscopists), followed by 20 endoscopist and 30 patient in-depth interviews, then an online questionnaire. Each stage will be thematically analysed to form the semi-structured questions for the next stage. The target population will be endoscopists who perform colonoscopy and people who have undergone, or refused to undergo, a colonoscopy. Focus groups will be performed in groups of 6-10 participants, and both interview and focus groups will be performed via video/teleconferencing.

ELIGIBILITY:
Inclusion Criteria:

One of:

* undergone a colonoscopy
* offered a colonoscopy but declined
* perform or training to perform colonoscopy

Exclusion Criteria:

* Non-English speaking
* Unable to comply with any study requirements
* New or ongoing diagnosis of bowel cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient invitations will be sent out to those on the emailing list of Crohns and Colitis UK, Bowel Cancer UK, Bowel Research UK and advertised on social media, to target populations likely to have experience in colonoscopy and across a variety of indications. Advertising posters will be placed in the outpatient and endoscopy departments of Leeds Teaching Hospitals NHS Trust.
  Endoscopist invitations will be via emailing lists to JAG and ACPGBI members, Gastroenterology trainees and nurse endoscopist groups and advertised on social media, attempting to get a representation of various specialties and roles involved in colonoscopy, such as Gastroenterologists (Consultants and trainees), Surgeons and non-medical endoscopists.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient participant reported experience of colonoscopy - focus group | 1 year
  Descriptive reporting on thematic analysis of a focus group involving patients exploring their experience of colonoscopy.
Patient participant reported experience of colonoscopy - interviews | 1 year
  Descriptive reporting on thematic analysis following interviews of patients exploring their experience of colonoscopy.
Patient participant reported barriers to colonoscopy - focus group | 1 year
  Descriptive reporting on thematic analysis following a focus groups involving patients exploring the barriers to colonoscopy.
Patient participant reported barriers to colonoscopy - interviews | 1 year
  Descriptive reporting on thematic analysis following interviews of patients exploring the barriers to colonoscopy.
Colonoscopist participant perceptions of the patient experience of colonoscopy - focus group | 1 year
  Descriptive reporting on thematic analysis of a focus groups involving colonoscopists exploring what they feel to be important patient experience measures in colonoscopy.
Colonoscopist participant perceptions of the patient experience of colonoscopy - interviews | 1 year
  Descriptive reporting on thematic analysis of interviews of colonoscopists exploring what they feel to be important patient experience measures in colonoscopy.
Colonoscopist participant perceptions of the patient barriers to colonoscopy - focus group | 1 year
  Descriptive reporting on thematic analysis of a focus group involving colonoscopists exploring what they feel to be important barriers to colonoscopy for patients.
Colonoscopist participant perceptions of the patient barriers to colonoscopy - interviews | 1 year
  Descriptive reporting on thematic analysis of interviews of colonoscopists exploring what they feel to be important barriers to colonoscopy for patients.
PREMs patient participant questionnaire | 1 year
  Level of importance given to the reported patient experience measures and barriers (as developed from the interviews and focus groups), assessed by Likert style questions.
PREMs colonoscopist participant questionnaire | 1 year
  Perceived level of importance given to the reported patient experience measures and barriers (as developed from the interviews and focus groups), assessed by Likert style questions.

SECONDARY OUTCOMES:
Patient participants thoughts and feelings about robotic colonoscopy - focus group | 1 year
  Descriptive reporting following thematic analysis of a focus group exploring patients' thoughts and feeling on a new colonoscopy technology - a magnetic robotic colonoscope.
Patient participants thoughts and feelings about robotic colonoscopy - interview | 1 year
  Descriptive reporting following thematic analysis of interviews exploring patients' thoughts and feeling on a new colonoscopy technology - a magnetic robotic colonoscope.
Patient participants thoughts and feelings about artificial intelligence - focus group | 1 year
  Descriptive reporting following thematic analysis of a focus group exploring patients' thoughts and feeling on a artificial intelligence in endoscopy
Patient participants thoughts and feelings about artificial intelligence - interviews | 1 year
  Descriptive reporting following thematic analysis of interviews exploring patients' thoughts and feeling on a artificial intelligence in endoscopy
Colonoscopist participants thoughts and feelings about robotic colonoscopy - focus group | 1 year
  Descriptive reporting following thematic analysis of a focus group exploring colonoscopists' thoughts and feeling on a new colonoscopy technology - a magnetic robotic colonoscope.
Colonoscopist participants thoughts and feelings about robotic colonoscopy - interviews | 1 year
  Descriptive reporting following thematic analysis of interviews exploring colonoscopists' thoughts and feeling on a new colonoscopy technology - a magnetic robotic colonoscope.
Colonoscopist participants thoughts and feelings about artificial intelligence - focus groups | 1 year
  Descriptive reporting following thematic analysis of a focus group exploring colonoscopists' thoughts and feeling on a artificial intelligence in endoscopy.
Colonoscopist participants thoughts and feelings about artificial intelligence - interviews | 1 year
  Descriptive reporting following thematic analysis of interviews exploring colonoscopists' thoughts and feeling on a artificial intelligence in endoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
If possible to suitably anonymise, exerts from the focus group and interview transcripts will be made available.